CLINICAL TRIAL: NCT04539886
Title: A Multicenter, Prospective, Randomized, Comparison IDE Study Between the Pulse Biosciences CellFX System and Electrodessication (Hyfrecator Electrosurgical) for the Treatment of Sebaceous Hyperplasia (SH) Lesions
Brief Title: Comparative Study Between CellFX and Electrodessication in Sebaceous Hyperplasia (SH) Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP-SC-012
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Skin Lesion; Skin Abnormalities; Sebaceous Hyperplasia
Keywords: CellFX; Nano-Pulse Stimulation; NPS; Clearance
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receiving the two treatments in a split-face design with CellFX being used on only one side of the face and Electrodessication on the other side. The randomization assignment will include the type of treatment and which side of the face.
Who Masked: Outcomes Assessor
Masking Description: The Principal Investigator will select a sub investigator to be the blinded investigator to classify healing characteristics and aesthetic appearance of each subject's selected lesions at baseline and treated lesions post treatment and at 7-days, 30-days, and 60-days following the last CellFX treatment or Electrodessication. This sub investigator will be blinded to the treatment assignment. The subject may not be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- CellFX System (Experimental): The CellFX System consists of a electrical pulse console combined with a handpiece coupled with a sterile single patient-use treatment tip (1.5 x 1.5mm, 2.5 x 2.5mm, and 5.0 x 5.0mm). Based on the size of the SH lesion and treatment tip used, a predetermined treatment energy setting is selected to deliver a sequence of electrical pulses to the SH lesion area directly beneath the treatment tip.
  Interventions: Device: CellFX System
- Intralesional Electrodesiccation (Active Comparator): Intralesional Electrodesiccation involves using a Hyfrecator electrosurgical unit and a non-insulated epilation needle electrode to apply a high-frequency electric current within the lesion.
  Interventions: Device: Intralesional Electrodesiccation

INTERVENTIONS:
Device: CellFX System — CellFX System consists of a console combined with a handpiece and coupled with a sterile single patient-use treatment tip (1.5 x 1.5mm, 2.5 x 2.5mm, and 5.0 x 5.0mm)
  Arms: CellFX System
Device: Intralesional Electrodesiccation — Hyfrecator electrosurgical unit with a non-insulated needle-shaped electrode
  Arms: Intralesional Electrodesiccation

SUMMARY:
This study is designed as a multi-center, single-blinded, prospective, randomized, study to compare the safety and effectiveness of the CellFX System to the comparator group, Electrodessication for the treatment of SH lesions in healthy adult subjects.

DETAILED DESCRIPTION:
This SH comparative study will evaluate safety and efficacy in a split face design using the CellFX System and pre-defined energy profile for all primary and secondary treatments based on Fitzpatrick Skin Types and tip size. The comparator group will be treated with the same standardized intralesional electrodesiccation procedure conducted by all participating clinical sites. Subjects with 4-10 qualifying SH lesions on the face except the scalp, nose and within the orbital region will be enrolled. Each subject will be evaluated by the blinded site investigator at 7-days, 30-days, and 60-days post-initial CellFX and Electrodessication treatments. At the 30-day follow-up visit, lesions will be evaluate using Global Aesthetic Improvement Scale (GAIS), for eligibility to receive an additional treatment. In case of a second treatment, the subject will be evaluated by the blinded site investigator at 30-days and 60-days post-retreatment. Photography of the study lesions will be captured along with the blinded site investigator assessments at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 21 and no older than 80 years of age.
* Subject gives voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subject must comply with study procedures including follow-up visits.
* Subject is willing to have SH lesions treated in a single treatment session and understands that their lesion(s) may undergo a second treatment session at a subsequent visit.
* Subject must have a minimum of four SH lesions and up to 10 SH lesions to be treated and the subject must have at least two SH lesions located on each side of the face.
* For study purposes, the SH lesions must be no greater than 2 mm in height and must not exceed 5 mm x 5 mm at their largest dimension. The subject's lesions cannot be located within the eye orbit, nose, or scalp.
* Subject consents to have photographs taken of the SH lesion(s).
* Subject agrees to refrain from using all other lesion removal products or treatments (e.g. retinols, retinoids, and exfoliating products) to the treated SH lesions or any new SH lesions during the study period.
* Subject agrees to refrain from prolonged sun exposure during the study period.

Exclusion Criteria:

* Subject has an implantable electronic medical device.(i.e., pacemaker, implantable cardioverter defibrillator)
* Subject has an active infection or history of infection in designated test area within 90 days prior to first treatment.
* Subject is not willing or able to sign the Informed Consent.
* Subject is known to be immune compromised.
* Subject is prone to developing hypertrophic scars or to be a keloid producer.
* Subject has allergies to Lidocaine or Lidocaine-like products.
* Subject is employed by the sponsor, clinic site, or entity associated with the conduct of the study.
* Have any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study.
* Use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study.
* Subject was previously treated with CellFX for SH lesions.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (5):
- United States (5):
  - Investigate MD, LLC, Scottsdale, Arizona
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - Dermatology, Laser & Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina
  - Austin Institute for Clinical Research, Inc., Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a prospective, randomized, single-blinded, split-face design in a total of 60 participants with a minimum of 4 and a maximum of 10 SH lesions.
Pre-assignment Details: Not applicable, since randomization occurred at the time of enrollment, defined as the time when intervention of the device occurred.
Units Other Than Participants: SH Lesions
Groups:
- Participants Treated With CellFX System: The CellFX System consists of an electrical pulse console (similar to devices used to electro-coagulate tissue) combined with a handpiece which is held by the clinician during application of pulses directly to the skin surface. The handpiece is coupled to a sterile, single patient-use non-insulated treatment tip. Once the electrical pulse console is turned on and a predetermined treatment energy setting is selected, a sequence of preprogrammed electrical pulses is administered to an area of skin directly beneath the treatment tip.
- Participants Treated With Intralesional Electrodessication: Intralesional Electrodessication involves using a Hyfrecator electrosurgical unit and a non-insulated epilation needle electrode to apply a high-frequency electric current within the lesion.
  Intralesional Electrodessication: Hyfrecator electrosurgical unit with a non-insulated needle-shaped electrode
Period: Overall Study
Arm/Group | Participants Treated With CellFX System | Participants Treated With Intralesional Electrodessication
Started | 60; 188 SH Lesions (Design was a split-face design, so all 60 participants are in each arm, however the total number of SH lesions are defined by type of treatment.) | 60; 190 SH Lesions (Design was a split-face design, so all 60 participants are in each arm, however the total number of SH lesions are defined by type of treatment.)
Completed | 60; 187 SH Lesions | 60; 189 SH Lesions
Not Completed | 0; 1 SH Lesions | 0; 1 SH Lesions

BASELINE CHARACTERISTICS:
Population: The Study Design was a split-face design, so all 60 participants are presented in the baseline analysis population.
Groups:
- All Participants: All participants received prospective, randomized, single-blinded treatments using the CellFX System and Intralesional Electrodessication in a split-face study design. Participants were randomized to receive an initial treatment and a possible secondary treatment at 30 days with either the CellFX System on 1 side of the face and electrodessication on the other side.
  The CellFX System consists of an electrical pulse console (similar to devices used to electro-coagulate tissue) combined with a handpiece which is held by the clinician during application of pulses to the skin surface. The handpiece is coupled to a sterile, single patient-use non-insulated treatment tip. Once the electrical pulse console is turned on and a predetermined treatment energy setting is selected, a sequence of preprogrammed electrical pulses is administered to an area of skin directly beneath the treatment tip.
  The active comparator was electrodessication using the Hyfrecator electrosurgical unit with a non-insulated needle-shaped tip.
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 2
  Unknown or Not Reported | 2
Fitzpatrick Skin Type Class [Count of Participants; unit: Participants]
  Class II | 46
  Class III | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lesions With Improvement as Assessed With the Global Aesthetic Improvement Scale (GAIS)
Description: Percentage of SH Lesions with Improvement as Assessed by Blinded Investigator During Live Assessments based on Global Aesthetic Improvement Scale (GAIS). The Global Aesthetic Improvement Scale ranges from 1=Very Much Improved or Excellent Corrective Result to 5=Worsened Appearance Compared with Original Condition. The primary effectiveness endpoint of improvement at 60-days post-last treatment as assessed "live" by the blinded site investigator using the 5-point GAIS
Time Frame: 60 days post last CellFX or Electrodessication treatment, up to a maximum of 3 months.
Population: 2.5mm SH lesions were assessed at 60-days post-last treatment of the lesion with either CellFX or Electrodessication by blinded Investigator during live assessments using Global Aesthetic Improvement Scale (GAIS). The Global Aesthetic Improvement Scale ranges from 1=Very Much Improved or Excellent Corrective Result to 5=Worsened Appearance Compared with Original Condition.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Participants Treated With CellFX System | Participants Treated With Intralesional Electrodessication
Number analyzed (Participants) | 59 | 59
Number analyzed (Lesions) | 121 | 106
percentage of lesions | 76.2 [67.0 to 85.5] | 75.5 [66.6 to 84.4]

2. Primary Outcome: Percentage of Lesions With Hyperpigmentation, Hypopigmentation and Scarring as Assessed by Blinded Investigator During Live Assessments
Description: The first co-primary safety endpoint includes the percentage of lesions showing hyperpigmentation and scarring as assessed by the blinded Investigator at 60 days after the last treatment with CellFX or Electrodessication
Time Frame: 60 days post last CellFX or Electrodessication treatment, up to a maximum of 3 months.
Population: Subjects with 2.5mm lesions
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Participants Treated With CellFX System | Participants Treated With Intralesional Electrodessication
Number analyzed (Participants) | 59 | 59
Number analyzed (lesions) | 120 | 107
percentage of lesions | 15.1 [7.68 to 22.40] | 11.1 [5.19 to 17.0]

3. Primary Outcome: Percentage of Lesions With Skin Textual Changes as Assessed by Blinded Investigator During Live Skin Assessment
Description: The second co-primary safety endpoint of skin textural changes including; flaking, erythema, crusting, scabbing, or other skin irregularities was assessed by the blinded site investigator at 30 days post last CellFX or Electrodessication treatment.
Time Frame: 30 days post last CellFX or Electrodessication treatment, up to a maximum of 2 months
Population: Subjects with 2.5mm lesions with Pre-specified safety margin (95% CIU<15%)
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Participants Treated With CellFX System | Participants Treated With Intralesional Electrodessication
Number analyzed (Participants) | 59 | 59
Number analyzed (lesions) | 118 | 107
percentage of lesions | 6.87 [2.12 to 11.6] | 10.2 [3.84 to 16.6]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 6 months
Description: Percent of non-serious AEs are reported per participants
Groups:
- Participants Treated With CellFX System: The CellFX System consists of a electrical pulse console combined with a handpiece coupled with a sterile single patient-use treatment tip (1.5 x 1.5mm, 2.5 x 2.5mm, and 5.0 x 5.0mm). Based on the size of the SH lesion and treatment tip used, a predetermined treatment energy setting is selected to deliver a sequence of electrical pulses to the SH lesion area directly beneath the treatment tip.
  CellFX System: CellFX System consists of a console combined with a handpiece and coupled with a sterile single patient-use treatment tip (1.5 x 1.5mm, 2.5 x 2.5mm, and 5.0 x 5.0mm)
- Participants Treated With Intralesional Electrodesiccation: Intralesional Electrodesiccation involves using a Hyfrecator electrosurgical unit and a non-insulated epilation needle electrode to apply a high-frequency electric current within the lesion.
  Intralesional Electrodesiccation: Hyfrecator electrosurgical unit with a non-insulated needle-shaped electrode
Arm/Group | Participants Treated With CellFX System | Participants Treated With Intralesional Electrodesiccation
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 3/59 | 0/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With CellFX System (N=59) | Participants Treated With Intralesional Electrodesiccation (N=59)
Swelling (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — Mild swelling at site of lesion treatment that resolved within 7 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04539886/Prot_SAP_000.pdf